CLINICAL TRIAL: NCT05953441
Title: Artificial Intelligence Versus Human-controlled Doctor in Virtual Reality Simulation for Sepsis Team Training: Randomized Controlled Trial
Brief Title: Artificial Intelligence Versus Human-controlled Doctor in Virtual Reality Simulation for Sepsis Team Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Ministry of Education, Singapore (Other Government)
Responsible Party: Principal Investigator, Liaw Sok Ying, Assoc Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NUS-IRB-2022-202
Record Dates: First submitted 2023-07-10; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Sepsis
Keywords: artificial intelligence; team training; virtual reality simulation; health care education
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: Prospective 2-arm randomized controlled trial with a pretest-posttest study design
Who Masked: Outcomes Assessor
Masking Description: The simulation-based assessment videos were sent for rating by 2 assessors, who were blinded to the groupings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-powered group (Experimental): Participants participated in a 2-hour Virtual Reality Simulation (VRS), which consisted of 2 simulation scenarios. Participants had to perform nursing assessment and management of virtual patient, followed by communicating with an AI virtual doctor.
  Interventions: Other: AI-powered doctor
- Human-controlled group (Active Comparator): Participants participated in a 2-hour Virtual Reality Simulation (VRS), which consisted of 2 simulation scenarios. Participants had to perform nursing assessment and management of virtual patient, followed by communicating with a doctor avatar controlled by the medical student.
  Interventions: Other: Human-controlled doctor avatar

INTERVENTIONS:
Other: AI-powered doctor — AI-powered virtual doctor
  Arms: AI-powered group
Other: Human-controlled doctor avatar — Virtual doctor avatar controlled by the medical student.
  Arms: Human-controlled group

SUMMARY:
The purpose of the study is to compare the effectiveness of Artificial Intelligence virtual doctor with human-controlled virtual doctor avatars on nursing students' sepsis care and interprofessional communication.

ELIGIBILITY:
Inclusion Criteria:

1. All Year 3 NUS nursing students in Academic Year 2022
2. Individuals 20 years old and above; and
3. Consent to be video and/or audio-recorded

Exclusion Criteria:

1. Year 1, 2 and 4 NUS nursing students;
2. Incapable of giving informed consent;
3. Unable to understand and/or speak in English language;
4. Have visual, speech, and/or hearing impairment; and
5. Do not agree to be video and/or audio-recorded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-11-13 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Sepsis Knowledge on the 18-item sepsis knowledge test immediately after interventions. | Baseline and immediately after 2-hour VRS
  The 8-item communication knowledge and 18-item sepsis knowledge tests were developed and content validated by a multidisciplinary team comprising a medical doctor, an advanced practice nurse, and nursing academics.

SECONDARY OUTCOMES:
Change from Baseline in Team Communication Knowledge on the 8-item communication knowledge test immediately after interventions. | Baseline and immediately after 2-hour VRS
  The 8-item communication knowledge and 18-item sepsis knowledge tests were developed and content validated by a multidisciplinary team comprising a medical doctor, an advanced practice nurse, and nursing academics.
Change from Baseline in Team Communication Self-Efficacy on the 6-item Patient Clinical Information Exchange and Interprofessional Communication Self-Efficacy Scale immediately after interventions. | Baseline and immediately after 2-hour VRS
  The Patient Clinical Information Exchange and Interprofessional Communication Self-Efficacy Scale is a validated and self-reported instrument using a 0-100 Likert scale, which measures participants' perceptions of self-efficacy in team communication based on the ISBAR communication strategy.
Sepsis Care Performance through a 15-minute video-recorded simulation-based assessment within 2 weeks of postintervention. | Within 2 weeks of postintervention.
  2 independent raters used the validated RAPIDS (Rescuing A Patient In Deteriorating Situation) tool to measure nurses' simulation performance in assessing and managing a deteriorating patient.
Team Communication Performance through a 15-minute video-recorded simulation-based assessment within 2 weeks of postintervention. | Within 2 weeks of postintervention.
  2 independent raters used a validated 9-item team communication scale to assess nurses' simulation performance in communicating with doctor using the TeamSTEPPS communication strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Sok Ying Liaw, Principal Investigator — National University of Singapore
Locations (1):
- Alice Lee Centre for Nursing Studies, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
The data sets collected or analyzed during the study are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Liaw SY, Tan JZ, Bin Rusli KD, Ratan R, Zhou W, Lim S, Lau TC, Seah B, Chua WL. Artificial Intelligence Versus Human-Controlled Doctor in Virtual Reality Simulation for Sepsis Team Training: Randomized Controlled Study. J Med Internet Res. 2023 Jul 26;25:e47748. doi: 10.2196/47748. PMID 37494112